CLINICAL TRIAL: NCT00671606
Title: Hysteroscopic Injection of Tracers for Sentinel Node Identification in Women With Endometrial Cancer
Brief Title: Hysteroscopic Lymphatic Mapping for Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-0206
Record Dates: First submitted 2008-04-29; First posted 2008-05-05 (Estimated); Results first posted 2011-07-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2012-04

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Lymphatic Mapping; Sentinel Node Identification; Lymph Node; Intraoperative lymphatic mapping; Total hysterectomy; Bilateral salpingooophorectomy; Lymph node staging; Laparotomy; Laparoscopy
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative Lymphatic Mapping (Experimental): Intraoperative sentinel lymph node identification (lymphatic mapping)
  Interventions: Procedure: Intraoperative Lymphatic Mapping

INTERVENTIONS:
Procedure: Intraoperative Lymphatic Mapping — Intraoperative hysteroscopic injection of patent blue dye and radiocolloid for detection of sentinel lymph nodes.

SUMMARY:
The goal of this clinical research study is to learn if a procedure called intraoperative (during surgery) lymphatic mapping can be used to find the sentinel lymph node in patients with endometrial cancer.

DETAILED DESCRIPTION:
Experimental Procedures:

Lymph nodes are oval-shaped glands where immune reactions occur. For patients with endometrial cancer, lymph node status is an important factor for planning the cancer treatment course and predicting the status of the cancer. The "sentinel" node is the lymph node closest to the main tumor area, and it is believed to be at greatest risk for spread of the cancer. If the sentinel node does not contain cancer cells, then the remaining lymph nodes are usually cancer-free.

In this study, researchers want to study possibly using lymphatic mapping in future patients as an alternative to completely removing the lymph nodes in the pelvis (hip area) and para-aortic (upper abdomen) area.

Intraoperative sentinel lymph node identification (lymphatic mapping) uses 2 techniques. The first technique involves injecting a small amount of weak radioactive material, and the second involves injecting a drug called isosulfan blue or methylene blue. These techniques are being studied to see if the surgeon can locate ("map") lymph nodes that may contain tumor cells.

Routine Surgical Treatment:

As part of routine care, all participants in this study will have surgery to remove the uterus, cervix, 1-2 inches of the vagina, fallopian tubes, ovaries, and the lymph nodes in 2 areas of the waist.

Study Procedures:

If you agree to take part in this study, after you have been given the anesthetic for your surgery, your uterus will be examined to locate the tumor(s). After the tumor(s) are located, they will be injected with a radioactive substance called Tc-99m sulfur colloid. The tumors will then be injected with a dye called isosulfan blue or methylene blue, which is used to turn the sentinel node blue.

Before and during your surgery, a gamma counter (a special hand-held instrument that measures radioactivity) will be used to identify lymph nodes that have absorbed the Tc-99m sulfur colloid. The surgeon will also be able to see the lymph nodes that have absorbed the blue dye.

Information Collection:

In addition to the study procedures, researchers will collect clinical information about you that will be compared with the study results. This information includes your date of birth, age, race, height, weight, number of any past pregnancies and deliveries, any other medical conditions, and any earlier surgeries. It also includes the date of the cancer diagnosis, the status of the cancer diagnosis before surgery, the status of the disease, and the results of routine scans before surgery (chest x-ray and computed tomography [CT] or magnetic resonance imaging [MRI] scan, if performed).

Length of Study Participation:

Your participation in this study will be over after the 15-20 minute procedure for identifying the sentinel nodes. The routine surgery will occur after that, which can take up to 5 hours.

This is an investigational study. Tc-99m sulfur colloid, the blue dye (either isosulfan blue or methylene blue), and the gamma counter are FDA approved for the procedures used in this study.

Performing lymph node mapping and sentinel node identification during surgery in patients with endometrial cancer is considered experimental.

Up to 20 women will take part in this multicenter study. Up to 10 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy confirmed endometrial cancer who have been dispositioned to undergo total hysterectomy, bilateral salpingooophorectomy and lymph node staging.
2. Surgical procedures may be performed by either laparotomy or laparoscopy.
3. If computed tomography, magnetic resonance imaging, lymphangiography, or ultrasound has been performed for preoperative assessment, there must be no evidence of metastases. Imaging is not mandatory.
4. Patients who have signed an approved informed consent and authorization permitting release of personal health information.

Exclusion Criteria:

1. Patients with a preoperative diagnosis of grade I endometrioid adenocarcinoma of the uterus.
2. Patients with uterine papillary serous carcinoma.
3. Patients who have undergone endometrial ablation or a myomectomy within 1 year of the surgery for endometrial cancer.
4. Patients with known allergies to triphenylmethane compounds or technetium-99 radiocolloid.
5. Patients with a history of retroperitoneal surgery.
6. Patients with a history of pelvic radiation.
7. Patients with no lesion visible on hysteroscopy.
8. Patients with previous exposure to the tracer (to prevent risk of allergic reaction).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Frumovitz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - St. Luke's Episcopal Hospital, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 4/28/2008 to 5/4/2010. All participants were recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Intraoperative Lymphatic Mapping
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Lymphatic Mapping
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 56 [49 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Sentinel Node Identification Rate
Description: Feasibility of sentinel node identification rate using intraoperative hysteroscopic injection of patent blue dye and radiocolloid for the detection of sentinel lymph nodes in patients with endometrial cancer. Sentinel node identification before and during surgery using a gamma counter to identify lymph nodes that have absorbed Tc-99m sulfur colloid. Study feasibility assessed with enrollment of 20 participants, approximately 1 year.
Time Frame: 15-20 minute procedure prior to/during routine surgery for identifying the sentinel nodes
Population: Analysis was per protocol; no analysis conducted due to low detection rate.
Units Other Than Participants: Sentinel nodes
Arm/Group | Intraoperative Lymphatic Mapping
Number analyzed (Participants) | 0
Number analyzed (Sentinel nodes) | 0

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Intraoperative Lymphatic Mapping
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Early termination due to low detection rate of sentinel lymph nodes in the five participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No